CLINICAL TRIAL: NCT06555744
Title: A Phase 1, Open-label, Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Anti-tumor Activity of Ascending Doses of a Folate Receptor Alpha Antibody Drug Conjugate, ZW191, in Participants With Advanced Solid Tumors
Brief Title: A Study of ZW191 in Participants With Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zymeworks BC Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZWI-ZW191-101; 2024-512299-37-00 (EU CTIS Number)
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced or Metastatic Cancers; ADC; Folate alpha receptor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ZW191 (Experimental)
  Interventions: Drug: ZW191

INTERVENTIONS:
Drug: ZW191 — Administered intravenously

SUMMARY:
The purpose of this study is to find out if ZW191 is safe and can treat participants with advanced cancers, including ovarian, endometrial, and non-small cell lung cancers.

DETAILED DESCRIPTION:
Part 1 of the study will evaluate the safety and tolerability of ZW191. Part 2 of the study will further evaluate safety and explore the potential anti-tumor activity of ZW191.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically or cytologically confirmed diagnosis of cancers with evidence of locally advanced (unresectable), recurrent and/or metastatic disease.
* Measurable disease per RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
* Adequate cardiac function: Cardiac left ventricular function, as defined by left ventricular ejection fraction (LVEF) ≥ 50% as determined by either echocardiogram (ECHO) or multigated acquisition scan (MUGA).
* Other adequate organ function.

Exclusion Criteria:

* Known additional malignancy that is progressing or requires active treatment or may interfere with study endpoints.
* Has received prior Topoisomerase I inhibitor(TOPO1i) antibody drug conjugate treatment, regardless of washout period.
* Acute or chronic uncontrolled renal disease, pancreatitis, or liver disease.
* Severe chronic or active infections (including known active SARS-CoV-2 infection) requiring systemic therapy, including antibacterial, antifungal, or antiviral therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs; Part 1) | Up to 3 weeks
  Number of participants who experienced a DLT. DLTs include specifically defined adverse events (AEs) considered to be related to ZW191
Incidence of adverse events (AEs; Parts 1 and 2) | Up to approximately 2 years
  Number of participants who experienced AEs, adverse events of special interest (AESIs), or serious adverse events (SAEs)
Incidence of clinical laboratory abnormalities (Parts 1 and 2) | Up to approximately 2 years
  Number of participants who experienced a maximum severity of Grade 3 or higher post-baseline laboratory abnormality, including either hematology or chemistry. Grades are defined using National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE), version 5.0
Confirmed objective response rate (Part 2) | Up to approximately 2 years
  Number of participants who achieved a best overall response of either confirmed complete response (CR) or partial response (PR) during treatment according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

SECONDARY OUTCOMES:
Confirmed objective response rate (Part 1) | Up to approximately 2 years
  Number of participants who achieved a best overall response of either confirmed CR or PR during treatment according to RECIST v1.1
Clinical benefit rate (Parts 1 and 2) | Up to approximately 2 years
  Number of participants who achieved a best response of CR, PR, non-CR/non-progressive disease (PD), or stable disease (SD) lasting at least 180 days per RECIST v1.1
Duration of response (DOR; Part 2) | Up to approximately 2 years
  The time from the first objective response (CR or PR) to the first documented PD per RECIST v1.1 or death within 30 days of last dose of study treatment from any cause. Only participants who achieve a confirmed response will be included in the analysis
Disease control rate (DCR; Part 2) | Up to approximately 2 years
  Number of participants who achieved a best response of CR, PR, non-CR/non-PD (for participants who have only non-target lesions), or SD during treatment per RECIST v1.1
Progression-free survival (PFS; Part 2) | Up to approximately 2 years
  The time from the first dose of study treatment to the date of first documented PD per RECIST v1.1 or death from any cause
Best overall response (BOR; Part 2) | Up to approximately 2 years
Serum or plasma concentration and PK parameters of ZW191 (Parts 1 and 2) | Up to approximately 2 years
  Maximum serum concentration and trough concentration of ZW191
Incidence of anti-drug antibodies (ADAs; Parts 1 and 2) | Up to approximately 2 years
  Number of participants who develop ADAs

CONTACTS AND LOCATIONS:
Overall Officials: Akira Kojima, MD, Study Director — Zymeworks BC Inc.
Locations (24):
- United States (5):
  - Yale University, New Haven, Connecticut
  - The Arthur G. James Cancer Hospital and Richard J. Solove Research Institute, Columbus, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - NEXT Oncology, San Antonio, Texas
  - NEXT Virginia, Fairfax, Virginia
- Australia (2):
  - Linear Clinical Research, Nedlands
  - Royal North Shore Hospital Northern Sydney Cancer Centre, St Leonards
- Japan (4):
  - National Cancer Center Hospital East, Kashiwa-shi
  - Saitama Medical University International Medical Center, Saitama
  - National Cancer Center Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
- Singapore (3):
  - National University Health System (NUHS) - National University Cancer Institute Singapore (NCIS), Singapore
  - National Cancer Centre Singapore, Singapore
  - Curie Oncology, Singapore
- South Korea (7):
  - National Cancer Center, Goyang-si
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
- Spain (3):
  - Hospital Universitario Reina Sofia, Córdoba
  - Fundacion Instituto Valenciano de Oncologia (IVO), Valencia
  - Hospital Clinico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No